CLINICAL TRIAL: NCT06913010
Title: The Service Regulation DV 100 as an Organizational Structure for Establishing the Hospital Incident Command System
Brief Title: DV 100 as a Framework for the Hospital Incident Command System
Acronym: OrAKEL
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Prof. Erik Popp, MD (Unknown); Prof. Markus Ries, MD, PhD, MHSc, MA, FCP, FIBODM (Unknown); Janna Küllenberg, PhD (Unknown); Kirsten Bikowski (Unknown); Hanne Schäfer, RN, BS, MS (Unknown)
Responsible Party: Principal Investigator, Maik von der Forst, Deputy Medical Director of the Crisis and Disaster Management Unit, University Hospital Heidelberg
Other Study IDs: OrAKEL
Record Dates: First submitted 2025-03-25; First posted 2025-04-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Disaster; Crisis Response Plan; Emergency; Communication
Keywords: Hospital Incident Command System; Continental Staff System; Service Regulation DV 100; Disaster Management; Emergency Planning; Hospital Alarm and Emergency Planning; Organizational Structure; Crisis Management; Communication Processes; Transition Processes; Healthcare Emergency Response; Civil Protection; Disaster Assistance; Incident Command Structure; Emergency Management Systems
MeSH Terms: conditions — Emergencies; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- University Hospital Heidelberg staff eligible for deployment in the hospital incident command system: Only adult employees capable of giving informed consent are included. The study population comprises all University Hospital Heidelberg staff potentially involved in the hospital incident command system.
  Interventions: Other: No interventions.

INTERVENTIONS:
Other: No interventions. — This is an observational study with no interventions.

SUMMARY:
There is limited scientific research on the organizational structure of the Hospital Incident Command System. The Hospital Alarm and Emergency Planning manual by the German Federal Office of Civil Protection and Disaster Assistance (BBK) recommends a continental staff system-based organization, as outlined in the Service Regulation DV 100, similar to military, fire, and police structures. This approach is frequently discussed at professional conferences, but evidence on its functionality in hospitals is lacking. This study aims to generate new insights into the use of a continental staff system-based Hospital Incident Command System and qualitatively analyze transition and communication processes within the command structure.

ELIGIBILITY:
Inclusion Criteria:

* Participation in at least one hospital incident command system (ICS) training and, if applicable, in a ICS exercise.

Written informed consent from the employee for participation in the second part of the study (semi-structured interview)

Exclusion Criteria:

* Decline of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises all Heidelberg University Hospital staff potentially involved in the hospital incident command system
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Exploration of leadership communication and dynamics during the transition from routine clinical operations to an emergency situation | During the table-top exercise on May 26 and May 27, 2025.
  Assessed through semi-structured interviews based on Grounded Theory, a systematic method for developing theories through the analysis of qualitative data
Assessment of training and exercise effects within a structured (according to DV-100) hospital incident command system, including challenges, resistance, benefits, subjective participant experiences, potential improvements, and alternatives | During the table-top exercise on May 26 and May 27, 2025.
  Assessed through semi-structured interviews based on Grounded Theory, a systematic method for developing theories through the analysis of qualitative data

SECONDARY OUTCOMES:
Examination of the applicability of the traditional incident command concept in hospitals, considering a workforce largely inexperienced in continental staff system-based work. | During the table-top exercise on May 26 and May 27, 2025.
  Assessed through semi-structured interviews based on Grounded Theory, a systematic method for developing theories through the analysis of qualitative data
Evaluation of participants' operational confidence | During the table-top exercise on May 26 and May 27, 2025.
  Assessed through semi-structured interviews based on Grounded Theory, a systematic method for developing theories through the analysis of qualitative data
Analysis of communication behaviors within the command functions | During the table-top exercise on May 26 and May 27, 2025.
  Assessed through semi-structured interviews based on Grounded Theory, a systematic method for developing theories through the analysis of qualitative data
Assessment of the advantages and disadvantages of a structured hospital incident command system | During the table-top exercise on May 26 and May 27, 2025.
  Assessed through semi-structured interviews based on Grounded Theory, a systematic method for developing theories through the analysis of qualitative data

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes